CLINICAL TRIAL: NCT00008034
Title: A Phase I Study Of Cyclophoshamide And Epirubicin In Combination With Capecitabine (XELODA) (CEX) As Primary Treatment Of Locally Advanced/Inflammatory Or Large Operable Breast Cancer
Brief Title: Combination Chemotherapy Before Surgery in Treating Women With Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: EORTC-10991; EORTC-10991; IDBBC-10991-CEX
Record Dates: First submitted 2001-01-06; First posted 2004-02-03 (Estimated); Last update posted 2012-07-18 (Estimated); Status verified 2012-07

CONDITIONS: Breast Cancer
Keywords: stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; inflammatory breast cancer
MeSH Terms: conditions — Breast Neoplasms; Inflammatory Breast Neoplasms | interventions — Capecitabine; Cyclophosphamide; Epirubicin

INTERVENTIONS:
Drug: capecitabine
Drug: cyclophosphamide
Drug: epirubicin hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells and shrink tumors so they can be removed during surgery.

PURPOSE: Phase I trial to study the effectiveness of combination chemotherapy before surgery in treating women who have locally advanced, inflammatory, or large surgically removable breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the toxicity of neoadjuvant capecitabine, cyclophosphamide, and epirubicin in women with locally advanced or inflammatory or large operable breast cancer. II. Determine the maximum tolerated dose of this regimen in this patient population.

OUTLINE: This is a multicenter dose escalation study of capecitabine. Patients receive neoadjuvant cyclophosphamide IV and epirubicin IV on day 1 and oral capecitabine twice daily on days 1-14. Treatment continues every 21 days for a maximum of 6 courses in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of capecitabine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose limiting toxicity.

PROJECTED ACCRUAL: A total of 3-33 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed carcinoma of the breast Locally advanced or inflammatory disease (T4, any N or any T, N2 or N3 or T4d) OR Large operable disease (large T2 or T3 for which tumor shrinkage is needed) No distant metastasis on chest x-ray, liver ultrasound, or bone scan except for ipsilateral supraclavicular nodes No abnormal bone scintigrams that cannot be confirmed as benign Hormone Receptor Status Not specified

PATIENT CHARACTERISTICS: Age: 18 to 70 Sex: Female Menopausal status: Not specified Performance status: WHO 0-1 Life expectancy: Not specified Hematopoietic: Neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.25 times upper limit of normal (ULN) SGOT no greater than 2 times ULN Renal: Creatinine no greater than 1.5 times ULN Cardiovascular: LVEF normal by echocardiography or MUGA Other: Not pregnant or nursing Fertile patients must use effective contraception No other serious uncontrolled illnesses No uncontrolled psychiatric or addictive disorders No other concurrent or prior malignancy within the past 5 years except adequately treated basal or squamous cell skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy Surgery: See Disease Characteristics

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2000-02; Primary Completion 2000-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Herve Bonnefoi, MD, Study Chair — Hopital Cantonal Universitaire de Geneve
Locations (1):
- Hopital Cantonal Universitaire de Geneva, Geneva, Switzerland